CLINICAL TRIAL: NCT00747292
Title: Randomised Controlled Trial Comparing the Effects of Epidural, Spinal and PCA in Patients Undergoing Laparoscopic Colectomy.
Brief Title: Peri-Operative Management of Patients Undergoing Laparoscopic Colorectal Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minimal Access Therapy Training Unit (Other)
Responsible Party: Bruce Levy, MATTU
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07/H1111/70
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: Neoplasm; Diverticular Disease; Analgesia
Keywords: laparoscopic; colon; analgesia; fluid optimised
MeSH Terms: conditions — Neoplasms; Diverticular Diseases; Agnosia | interventions — Injections, Epidural; Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Epidural (Active Comparator): Epidural
  Interventions: Procedure: epidural
- 2 (Active Comparator): Spinal
  Interventions: Procedure: Spinal
- 3 (Active Comparator): Patients in this limb receive a PCA
  Interventions: Procedure: PCA

INTERVENTIONS:
Procedure: epidural — Patients in this limb receive epidural analgesia
  Arms: Epidural
Procedure: PCA — Patients in this limb receive a PCA for their pain control
  Arms: 3
Procedure: Spinal — Patients in limb will receive spinal analgesia
  Arms: 2

SUMMARY:
The aim is to ascertain which method out of epidural, spinal or patient controlled analgesia (PCA) is the most appropriate in fluid optimised patients after laparoscopic colorectal surgery in terms of pain control, length of hospital stay and time for gut recovery. The second aim is to assess the physiological changes that occur when the patient is placed in steep trendelenberg position together with the creation of the pneumoperitoneum.

DETAILED DESCRIPTION:
Patients will be randomized into one of 3 groups - A, B or C. In order to remove the major confounding factor of hypovolaemia, all patients will have an oesophageal doppler inserted in order to achieve fluid optimisation. Each group will then either have an epidural, spinal or a PCA for post operative analgesia depending on the randomisation. All patients will follow a common postoperative care pathway to standardize the other factors.

Patients will be asked to report parameters including pain visual analogue score (VAS) chart three times a day. Recovery of bowel functions (passage of flatus, bowel movement, and diet intake), additional analgesia consumption, time to first ambulation, analgesia related side-effects and time to discharge will be recorded.

In addition whilst the patients fluid status is optimized during surgery with the oesophageal Doppler, the physiological changes that occur with the steep trendelenberg position and the pneumoperitoneum will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal disease that requires a bowel resection who agree to have laparoscopic surgery with placement of an oesophageal doppler and a central line and who agree to be randomised with regards to a post operative analgesic regime.

Exclusion Criteria:

* Patients will be excluded from the post operative analgesia trial if they have abnormal clotting, skin infection over or near the back, presence of neurological disorders or anatomical abnormalities of the vertebral column, or for a reason identified by the anaesthetist.
* Patients will also be excluded if there is a contra-indication to oesophageal doppler such as oesophageal disease, recent oesophageal or upper airway surgery, moderate to severe aortic valve disease and bleeding diathesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | Once the patient is safe to go home

SECONDARY OUTCOMES:
Pain, time till flatus, time till bowels open, incidence of nausea and vomiting, quality of life | Once secondary outcomes are successful, patient can go home

CONTACTS AND LOCATIONS:
Overall Officials: Tim Rockall, FRCS, Study Director — Minimal Access Therapy Training Unit
Locations (1):
- MATTU, Guildford, Surrey, United Kingdom

REFERENCES:
- [Background] Senagore AJ, Delaney CP, Mekhail N, Dugan A, Fazio VW. Randomized clinical trial comparing epidural anaesthesia and patient-controlled analgesia after laparoscopic segmental colectomy. Br J Surg. 2003 Oct;90(10):1195-9. doi: 10.1002/bjs.4223. PMID 14515286
- [Background] Senagore AJ, Whalley D, Delaney CP, Mekhail N, Duepree HJ, Fazio VW. Epidural anesthesia-analgesia shortens length of stay after laparoscopic segmental colectomy for benign pathology. Surgery. 2001 Jun;129(6):672-6. doi: 10.1067/msy.2001.114648. PMID 11391364
- [Background] Taqi A, Hong X, Mistraletti G, Stein B, Charlebois P, Carli F. Thoracic epidural analgesia facilitates the restoration of bowel function and dietary intake in patients undergoing laparoscopic colon resection using a traditional, nonaccelerated, perioperative care program. Surg Endosc. 2007 Feb;21(2):247-52. doi: 10.1007/s00464-006-0069-5. Epub 2006 Dec 9. PMID 17160649
- [Background] Kong SK, Onsiong SM, Chiu WK, Li MK. Use of intrathecal morphine for postoperative pain relief after elective laparoscopic colorectal surgery. Anaesthesia. 2002 Dec;57(12):1168-73. doi: 10.1046/j.1365-2044.2002.02873.x. PMID 12437707